CLINICAL TRIAL: NCT05651009
Title: Comparison of the in Vivo Stability of 2 Cementless TKA Designs Using CT Micromotion Analysis - A Randomized Controlled Trial
Brief Title: Comparison of the in Vivo Stability of 2 Cementless TKA Designs
Acronym: ClessTKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Oslo University Hospital (Other); Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 520246
Record Dates: First submitted 2022-11-23; First posted 2022-12-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: CT based micromotion analysis; CTMA; Cementless TKA; Uncemented TKA; Total knee replacement; Total knee arthroplasty; TKR; GMK Sphere; Tritanium
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Double blinded study (patient and research nurse)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Cementless Triathlon Tritanium 3D printed TKA
  Interventions: Procedure: TKA
- Study group (Experimental): GMK Sphere cementless 3D printed TKA
  Interventions: Procedure: TKA

INTERVENTIONS:
Procedure: TKA — Total knee artroplasty with medial parapatellar incision and mechanical alignment without navigation

SUMMARY:
The goal of this randomized controlled trial is to analyze the stability of a cementless Total Knee Arthroplasty (TKA) over time and compare it to a well-documented implant in patients with knee osteoarthritis. The main aim is to answer if there is a difference in stability over time as a measure of long time survivorship in these 2 implants.

50 participants will be randomly allocated to receive either the Triathlon Tritanium (Stryker) or the Global Medacta Knee Sphere (GMK Sphere, Medacta) 3D printed cementless TKAs.

DETAILED DESCRIPTION:
Total joint replacement is an efficacious treatment for osteoarthritis of hips and knees. Both TKA and Total Hip Artrhoplasties (THA) have excellent implant survivorship. However, patients' satisfaction is lower in TKA than THA. A possible cause of the discrepancy is the unnatural knee kinematics after TKA. Various implants designs have been developed to solve the problem. The most common fixation mode is cemented TKA with good survival up to 15 years. However, newer series in younger patients also have shown lasting survival with cementless implants (Nilsson KG, Prudhon JL). Among various different designs, the medially stabilized total knee, which are designed to reproduce natural knee kinematics with a medial ball-in-socked design, is a promising implant design (No authors listed). Dynamically the medial pivot knee performs more naturally (Bragonzoni L,Petersen ET) compared to other designs. Most data for this design is available only for the cemented version. Up to now there is no safety study performed that confirms the stability over time for this implant with cementless fixation.

In this study, the investigators will therefore analyze the in vivo stability of an uncemented TKA with a medially stabilized design, and compare it with a well-documented comparable implant. In order to do this, the investigators will use the CT based micromotion analysis (Broden C, Broden C). This study will contribute to the understanding of fixation and lead to safety to the patient.

ELIGIBILITY:
Inclusion Criteria:

• Patients referred to Kristiansund Hospital for primary total knee replacement surgery for osteoarthritis with Kellgren & Lawrence grade 3 or 4

Exclusion Criteria:

* Preoperative severe deformity (Hip-Knee-Ankle angle of >5 (valgus) or <-15 degrees (varus) on a full-length leg image at weight bearing
* Preoperative flexion contracture more than 15°
* Less than 50 and more than 75 years of age at the time of surgery
* Use of walking aids because of other musculoskeletal and neuromuscular problems
* Preoperative diagnosis other than osteoarthritis or avascular necrosis (e.g. rheumatoid arthritis, tumours)
* Revision arthroplasty
* Obesity with BMI>35 g/m2
* Lateral collateral ligament deficient knee
* Previous knee joint infection
* Cognitive dysfunction or severe psychiatric disorders.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2028-06-25 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
CTMA Maximum Total Translation | Up to 2 years
  The highest total translation on the implant at each time point
CTMA Maximum Total Translation | Up to 5 years
  The highest total translation on the implant at each time point

SECONDARY OUTCOMES:
CTMA Total rotation | Up to 2 years
  Center of mass and peripheral points (degrees)
CTMA Total rotation | Up to 5 years
  Center of mass and peripheral points (degrees)
CTMA Total translation | Up to 2 years
  Center of mass and peripheral points (millimeters)
CTMA Total translation | Up to 5 years
  Center of mass and peripheral points (millimeters)
The Forgotten Joint Score (FJS) | Up to 2 years
  Patient Reported Outcome Measure PROMs). 12 item likert scale with scores from 0-4 (0=never, 4= allways). Mean value is multiplied with 25 and the subtracted from 100. Maximum score i 100 (excellent), minimum score is 0 (worse).
The Forgotten Joint Score (FJS) | Up to 5 years
  Patient Reported Outcome Measure PROMs). 12 item likert scale with scores from 0-4 (0=never, 4= allways). Mean value is multiplied with 25 and the subtracted from 100. Maximum score i 100 (excellent), minimum score is 0 (worse).
The Knee injury and Osteoarthritis Outcome Score (KOOS) | Up to 2 years
  Patient Reported Outcome Measure (PROMs). KOOS consists of 5 subscales; Pain, other Symptoms, Activites of Daily Living (ADL), Sport and Recreation Function (Sport/Rec) and knee-related Quality of Life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale
The Knee injury and Osteoarthritis Outcome Score (KOOS) | Up to 5 years
  Patient Reported Outcome Measure (PROMs). KOOS consists of 5 subscales; Pain, other Symptoms, Activites of Daily Living (ADL), Sport and Recreation Function (Sport/Rec) and knee-related Quality of Life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale
Range of motion | Up to 2 years
  From full extension to full flexion (degrees)
Range of motion | Up to 5 years
  From full extension to full flexion (degrees)
HKA | Up to 2 years
  Hip knee ankle angle measured on X-ray (degrees). Deviation from 0 is either varus (-) or valgus (+)
HKA | Up to 5 years
  Hip knee ankle angle measured on X-ray (degrees). Deviation from 0 is either varus (-) or valgus (+)

OTHER OUTCOMES:
BMI | Preoperative
  Body mass index (kg/m2)
Operation time | Intraoperative
  Time used in minutes from skin incision to wound closure.
Axial alignment of the tibia | Up to 1 week postoperative
  Measured by Bergers method (degrees internal or extarnal rotation)

CONTACTS AND LOCATIONS:
Overall Officials: Frank-David Øhrn, MD, PhD, Study Director — Møre og Romsdal Hospital Trust; Stephan M Röhrl, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Kristiansund Hospital, Møre and Romsdal Hospital Trust, Kristiansund, Møre and Romsdal, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately following publication and 5 years
Access Criteria: Researchers that want access to data

REFERENCES:
- [Background] Nilsson KG, Henricson A, Norgren B, Dalen T. Uncemented HA-coated implant is the optimum fixation for TKA in the young patient. Clin Orthop Relat Res. 2006 Jul;448:129-39. doi: 10.1097/01.blo.0000224003.33260.74. PMID 16826107
- [Background] Prudhon JL, Verdier R. Cemented or cementless total knee arthroplasty? - Comparative results of 200 cases at a minimum follow-up of 11 years. SICOT J. 2017;3:70. doi: 10.1051/sicotj/2017046. Epub 2017 Dec 12. PMID 29232186
- [Background] No authors listed. Australian Orthopaedic Association National Joint Replacement Registry (AOANJRR). Hip, Knee & Shoulder Arthroplasty: 2020 Annual Report, Adelaide; AOA, 2021: https://aoanjrr.sahmri.com/documents/10180/712282/Hip%2C+Knee+%26+Shoulder+Arthroplasty/bb011aed-ca6c-2c5e-f1e1-39b4150bc693 (date assessed October 29 2022).
- [Background] Bragonzoni L, Marcheggiani Muccioli GM, Bontempi M, Roberti di Sarsina T, Cardinale U, Alesi D, Iacono F, Neri MP, Zaffagnini S. New design total knee arthroplasty shows medial pivoting movement under weight-bearing conditions. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1049-1056. doi: 10.1007/s00167-018-5243-5. Epub 2018 Oct 27. PMID 30368560
- [Background] Petersen ET, Rytter S, Koppens D, Dalsgaard J, Hansen TB, Andersen MS, Stilling M. Medial congruent polyethylene design show different tibiofemoral kinematics and enhanced congruency compared to a standard symmetrical cruciate retaining design for total knee arthroplasty-an in vivo randomized controlled study of gait using dynamic radiostereometry. Knee Surg Sports Traumatol Arthrosc. 2023 Mar;31(3):933-945. doi: 10.1007/s00167-022-07036-w. Epub 2022 Jul 9. PMID 35809105
- [Background] Broden C, Sandberg O, Olivecrona H, Emery R, Skoldenberg O. Precision of CT-based micromotion analysis is comparable to radiostereometry for early migration measurements in cemented acetabular cups. Acta Orthop. 2021 Aug;92(4):419-423. doi: 10.1080/17453674.2021.1906082. Epub 2021 Apr 6. PMID 33821746
- [Background] Broden C, Olivecrona H, Maguire GQ Jr, Noz ME, Zeleznik MP, Skoldenberg O. Accuracy and Precision of Three-Dimensional Low Dose CT Compared to Standard RSA in Acetabular Cups: An Experimental Study. Biomed Res Int. 2016;2016:5909741. doi: 10.1155/2016/5909741. Epub 2016 Jul 10. PMID 27478832